CLINICAL TRIAL: NCT01286870
Title: Continued Access Study of the Mentor Becker Expander/Breast Implant
Brief Title: Becker Continued Access Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor terminated
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1222CA-1208-01; Becker CA Study
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Breast Reconstruction
Keywords: Primary Breast Reconstruction
MeSH Terms: interventions — Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reconstruction (Other): The study population will consist of women aged 18 or over who are undergoing primary breast reconstruction.
  The Reconstruction cohort will include subjects with loss of breast tissue due to mastectomy, contralateral breast for post-reconstruction symmetry or subjects with deformities secondary to disease, malignancy, trauma, and congenital deformity. Subjects in this cohort cannot have been implanted with breast implants, but may have tissue expanders. A Becker implant is considered a tissue expander until the port and fill tube have been removed. Women who undergo surgery primarily for a mastopexy will not be part of the reconstruction cohort.
  Interventions: Device: Mentor Becker 25 Expander/Breast Implant; Device: Mentor Becker 50 Expander/Breast Implant

INTERVENTIONS:
Device: Mentor Becker 25 Expander/Breast Implant — The breast implant is comprised of the Becker implant and the injection dome/fill tube and has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The inner lumen can be gradually filled with saline over an extended period of time via the fill tube by injecting saline through the injection dome. Once expanded to the desired volume, the fill tube and injection dome are removed through a small incision under local anesthetic, and the prosthesis remains in position as a breast implant.
  The Becker 25 Expander/Breast Implant has a silicone gel volume of approximately 25% and saline volume of approximately 75%. The Becker Expander/Breast Implant is available in sizes 150 - 800cc.
Device: Mentor Becker 50 Expander/Breast Implant — The breast implant is comprised of the Becker implant and the injection dome/fill tube and has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The inner lumen can be gradually filled with saline over an extended period of time via the fill tube by injecting saline through the injection dome. Once expanded to the desired volume, the fill tube and injection dome are removed through a small incision under local anesthetic, and the prosthesis remains in position as a breast implant.
  The Becker 50 Expander/Breast Implant has a 50% gel volume and a 50% saline volume, so a 400cc implant would nominally have 200cc of saline and 200cc of silicone. The Becker 50 Expander/Breast Implant is available in sizes from 300 to 700cc.

SUMMARY:
While Core Becker patient follow-up is being completed this Continued Access Study is designed to enroll patients at a limited rate per month to allow for continued physician and patient experience with the device.

Up to 12 patients per month at sites across the United States will be enrolled in this research study. These patients will be implanted with the Becker 25 or Becker 50 Expander/Breast implant and monitored for 10 years for safety.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Pre-market Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A pre-market approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision subjects. Every subject implanted had to be part of an adjunct study, in addition to being offered participation in a registry of gel-filled breast implant subjects. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in an IDE clinical trial.

A PMA for Mentor's MemoryGel™ Silicone Gel-Filled breast implants (which did not include the Becker Expander/Breast Implants) was subsequently filed with FDA in December 2003, and approved in November 2006 (P030053). As a condition of approval of P030053, new enrollment in Mentor's Adjunct Study has ceased, and women no longer have access to the Becker Expander/Breast Implants.

The Mentor Becker Expander/Breast Implant was used throughout the United States during this time (since 1992) under the Mentor Adjunct Study to allow continued access to the device and to collect some safety information, however was not evaluated in the MemoryGel Core Study. The gel fill used in the MemoryGel implants is the same gel fill that is used for the Becker device.

This protocol describes the study design procedures and population for a Continued Access (CA) Study for the Mentor Becker 25 and 50 Expander/Breast implants. While Core Becker patient follow-up is being completed, this CA Study is designed to enroll patients at a limited rate per month to allow for continued physician experience with the device. The safety data obtained may be used to provide supplemental information to the PMA. It will be requested that this study be initiated and renewed every six months until a final decision is reached regarding the Becker PMA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is genetic female, 18 years of age or older
* A candidate for primary breast reconstruction for cancer, trauma, surgical loss of breast tissue due to mastectomy, malignancy, contralateral post-reconstruction symmetry, or congenital deformity, including asymmetry (see Section 6.0 for definition)
* Signs the Informed Consent
* Agrees to return device to Mentor if explant necessary
* Agrees to comply with follow-up procedures, including returning for all follow-up visits
* Patient is a US citizen with a Social Security Number and understands English

Exclusion Criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment.
* Been implanted with any silicone implant including breast implants (e.g. silicone artificial joints or facial implants)
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondylarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Implanted metal or metal devices, history of claustrophobia or other condition that would make a MRI scan prohibitive
* Physician is intending to use the device for tissue expansion only

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2014-03-04 (Actual); Study Completion 2014-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Walker, Principal Investigator — Binghamton, NY
Locations (1):
- Mentor Worldwide LLC, Santa Barbara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Becker CA Study was an open-label, multi-center study to provide continued physician and patient experience with the smooth Becker 25 and 50 Expander/Breast Implant. Subjects included women who required primary breast reconstruction.
Period: Overall Study
Arm/Group | Reconstruction
Started (September 22, 2008) | 11
Completed (February 28, 2014) | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reconstruction
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 10
  Race: Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety by Incidence, Severity, and Duration of Adverse Events
Time Frame: 4 Years
Population: The study was prematurely discontinued. The sample size was not large enough for statistical significance.
  Because only 11 subjects were enrolled in the Becker CA Study, demographic information and key safety information were listed by subject only and no formal summary tables were prepared.
Measure: Number; unit: Events
Arm/Group | Reconstruction
Number analyzed (Participants) | 11
Events
  Number of Adverse Events (AEs) | 33
  Mild AEs | 32
  Moderate AEs | 1
  Severe AEs | 0
  Ongoing AEs at end of trial | 6
  Resolved AEs | 27
  AE resolution the same day as AE onset | 5
  AE resolution in 1 week (1-7 days) | 12
  AE resolution in 2 weeks (8-14 days) | 1
  AE resolution in 2-4 weeks (15-30 days) | 3
  AE resolution in 1-3 months (30-90 days) | 3
  AE resolution over 3 months (90+ days) | 3

2. Primary Outcome: Safety by Method of Resolution of Adverse Events
Time Frame: 4 Years
Population: as for outcome 1
Measure: Number; unit: Procedures
Arm/Group | Reconstruction
Number analyzed (Participants) | 11
Procedures
  Re-operation Procedures Without Explantation | 16
  Re-operation Procedures With Explantation | 9

ADVERSE EVENTS:
Description: Ten of the 11 subjects in the CA Study had one or more postoperative complications. Severity was mild for all but 1 moderate case of infection and 2 moderate cases of Grade III capsular contracture
Arm/Group | Reconstruction
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 10/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reconstruction (N=11)
Delayed Wound Healing (General disorders) | 4
Grade III Capsular Contracture (General disorders) | 5
Infection (Infections and infestations) | 4
Wound Dehiscence (General disorders) | 1
Breast - Unacceptably High Sensitivity (Injury, poisoning and procedural complications) | 1
Excess Tissue/Dog Ear (Injury, poisoning and procedural complications) | 1
Grade IV Capsular Contracture (General disorders) | 1
Seroma (General disorders) | 1
Extrusion (General disorders) | 1
Wrinkling (Injury, poisoning and procedural complications) | 1
Nipple - Unacceptably High Sensitivity (Injury, poisoning and procedural complications) | 1
Asymmetry (Injury, poisoning and procedural complications) | 1
Irritation/Inflammation (Injury, poisoning and procedural complications) | 2
Hypertrophic Scarring (Injury, poisoning and procedural complications) | 1
Necrosis (Injury, poisoning and procedural complications) | 3
Swelling (Excessive) (Injury, poisoning and procedural complications) | 1
Size Change - Patient Request (General disorders) | 2
Grade II Capsular Contracture w/Surgical (Injury, poisoning and procedural complications) | 2

LIMITATIONS AND CAVEATS:
Because only 11 subjects were enrolled in the Becker CA Study, demographic information and key safety information were listed by subject only and no formal summary tables were prepared.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No